CLINICAL TRIAL: NCT01632956
Title: Developing Culturally-Tailored Information-Based Support Groups for Chinese Immigrants With Breast Cancer: A Pilot Study
Brief Title: Developing Culturally-Tailored Information-Based Support Groups for Chinese Immigrants With Breast Cancer
Status: Withdrawn | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Cancer Support Community (Unknown); CHARLES B WANG COMMUNITY HEALTH CENTER (Unknown); Queens Health Network (Other)
Responsible Party: Sponsor
Other Study IDs: 12-105
Record Dates: First submitted 2012-06-29; First posted 2012-07-04 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Chinese Immigrants With Breast Cancer
Keywords: Support Groups; Breast cancer; Mandarin speaking; 12-105
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- in-person support group: This is a 1 year pilot study of the feasibility of participation in both in-person and virtual information-based, culturally tailored support groups for Chinese breast cancer patients.
  Interventions: Behavioral: in-person support group
- virtual support group: This is a 1 year pilot study of the feasibility of participation in both in-person and virtual information-based, culturally tailored support groups for Chinese breast cancer patients.
  Interventions: Behavioral: virtual support group

INTERVENTIONS:
Behavioral: in-person support group — Each support group will consist of 12 sessions. Thirty-two breast cancer patients of Chinese descent will be recruited to participate in the support groups (16 in the inperson groups and 16 in the virtual groups).
  Groups: in-person support group
Behavioral: virtual support group — Each support group will consist of 12 sessions. Thirty-two breast cancer patients of Chinese descent will be recruited to participate in the support groups (16 in the inperson groups and 16 in the virtual groups).
  Groups: virtual support group

SUMMARY:
There are few breast cancer support groups that focus on the specific needs of Chinese women. The purpose of this study is to learn about two different ways of providing support groups to help women of Chinese descent cope with the difficulties of a diagnosis of breast cancer and its treatment. The investigators want to learn about how best to support Chinese women with breast cancer by providing two different types of groups: an in-person support group and a virtual (online/phone) support group.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Non-US born
* Resident in the US < 20 years
* Of Chinese descent
* Age 21 years through 80 years
* Language spoken: Mandarin
* Diagnosis of breast cancer within 3 months prior to recruitment

  *Not required that breast cancer is the patients' first and/or only cancer diagnosis
* Currently receiving cancer treatment;
* Will be living continuously in the US for the next year
* Has a telephone that he/she is willing to use for the study

Exclusion Criteria:

* Presence of cognitive impairment disorder (i.e., delirium or dementia) sufficient to preclude meaningful informed consent and/or data collection
* Another household member is already enrolled.
* Prior participation in a cancer support group

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment will be conducted by the MSKCC Research Study Assistant (RSA) with the assistance of the treatment team and community partners. Patients of MSKCC and QCC will be approached in clinic waiting rooms by the RSA. ACS Asian Initiatives and the Charles B Wang Community Health Center are referral sites for this study.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
feasibility | 1 year
  To pilot and evaluate the feasibility of information-based, culturally-tailored in-person and virtual support groups for Chinese patients with breast cancer. The feasibility of participation in the in-person and virtual support groups will be measured by documenting patient accrual to the pilot study and attendance at the support groups.

SECONDARY OUTCOMES:
To compare the impact of participation | 1 year
  in the in-person versus virtual support groups on quality of life (QOL), pain, psychosocial outcomes (distress, depression, anxiety, self-efficacy in coping with cancer), and perceived social support. These outcomes will be measured through a baseline and exit Outcomes Survey.
To assess satisfaction with the support groups | 1 year
  All participants will complete the Brief Support Group Survey at the end of each support meeting to assess satisfaction with and to provide feedback on the usefulness of the meeting and the information presented, ease of understanding and cultural appropriateness of the information, effectiveness of the facilitator, and suggestions for change or improvement.
To assess Internet use | 1 year
  among support group participants. All patients approached for study participation will complete the Screening Tool, which includes questions related to Internet use. The Screening Tool will be used for all eligible patients (patients refusing to participate will still be asked to complete the screening tool).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Leng, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Queens Cancer Center of Queens Hospital, Jamaica, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/